CLINICAL TRIAL: NCT03412266
Title: Reduced Intensity Conditioning Regimen for Low- and Intermediate-risk Myelodysplastic Syndrome Patients Receiving Haploidentical Hematopoietic Stem Cell Transplantation
Brief Title: RIC Regimen for Low- and Intermediate-risk MDS Receiving Haplo-HSCT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Xiao-Jun Huang, Director, Peking University People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RIC Haplo-MDS
Record Dates: First submitted 2018-01-21; First posted 2018-01-26 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Myelodysplastic Syndromes
Keywords: RIC regimen; MDS; haplo-HSCT; survival
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Cytarabine; Busulfan; Cyclophosphamide; fludarabine; Semustine; Antilymphocyte Serum

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RIC regimen (Other): Low- and intermediate MDS patients without identical sibling donor or unrelated donor would receive RIC haplo-HSCT.
  RIC preconditioning regimen consisted of cytarabine (2 g/m2/day, days -10 to -9), busulfan (3.2 mg/kg/day on days -8 to -6), cyclophosphamide (1.0 g/m2/day, days -5 to -4), fludarabine (30 mg/m-2/day, days -6 to -2), semustine (250 mg/m-2, day -3), and rabbit antithymocyte globulin (thymoglobulin, 2.5 mg/kg/d, days -5 to -2; Sanofi, France).
  Interventions: Drug: Cytarabine

INTERVENTIONS:
Drug: Cytarabine — RIC preconditioning regimen consisted of cytarabine (2 g/m2/day, days -10 to -9), busulfan (3.2 mg/kg/day on days -8 to -6), cyclophosphamide (1.0 g/m2/day, days -5 to -4), fludarabine (30 mg/m-2/day, days -6 to -2), semustine (250 mg/m-2, day -3), and rabbit antithymocyte globulin (thymoglobulin, 2.5 mg/kg/d, days -5 to -2; Sanofi, France).
  Other Names: busulfan; Cyclophosphamide; Fludarabine; Semustine; antithymocyte globulin

SUMMARY:
This study aimed to evaluate the efficacy of reduced intensity conditioning (RIC) regimen in low- and intermediate-risk myelodysplastic syndrome (MDS) patients who receive haploidentical hematopoietic stem cell transplantation (haplo-HSCT). Haplo-HSCT is an effective treatment option for MDS patients who did not have identical sibling donor (ISD) or unrelated donor (URD). However, post-transplant transplant-related mortality (TRM) is one of the major causes for transplant failure in MDS patients, and the risk of TRM for haplo-HSCT recipients was higher than that of ISD recipients. RIC regimen can decrease the risk of TRM for haplo-HSCT recipients; however, the risk for relapse may increase in these patients. Thus, RIC regimen may be more appropriate for low- and intermediate-risk MDS patients receiving haplo-HSCT. The study hypothesis: Using RIC haplo-HSCT regimen in patients with low- and risk MDS can reduce TRM and improve survival.

DETAILED DESCRIPTION:
RIC regimen was given for low and intermediate MDS patients who would receive haplo-HSCT. The primary end point was transplant-related mortality. The secondary end points were overall survival, disease-free survival, relapse, , graft-versus-host disease (GVHD), and infections. Following time is 1 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had low- and intermediate-risk MDS without ISD nor URD receiving haploidentical hematopoietic stem cell transplantation

Exclusion Criteria:

* Patients having ISD or URD; patients having high-risk MDS; patients with active infection; patients with poor compliance; patients with organ failure

Ages: 1 Year to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-02-01 (Actual); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
Transplant-related mortality | Participants will be followed for an expected average of 1 years
  Death without disease progression or relapse

CONTACTS AND LOCATIONS:
Overall Officials: Xiao-Jun Huang, Principal Investigator — Peking University Institute of Hematology
Locations (1):
- Peking University Institute of Hematology,Beijing, Beijing, Beijing Municipality, China